CLINICAL TRIAL: NCT05476107
Title: A Phase 1 Study in up to 2 Parts, to Assess the Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of AMT-126 in the Fasted State (in Part 1) and to Evaluate the In Vivo Performance of an AMT-126 Oral Tablet Through Pharmacoscintigraphic Assessment in the Fed and Fasted State (in Optional Part 2) in Healthy Male and Female Subjects
Brief Title: SAD Study to Assess the Safety, Tolerability, PK, and In-Vivo Performance of AMT-126 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Applied Molecular Transport (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AMT-126-001; 2020-005779-11 (EudraCT Number)
Record Dates: First submitted 2022-06-22; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Radioactivity

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either receive AMT-126 or placebo (Part 1), Radiolabeled tablet (Part 2)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded (Part 1), Open Label (Part 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AMT-126 (Experimental): oral AMT-126
  Interventions: Drug: AMT-126
- Placebo (Placebo Comparator): oral placebo
  Interventions: Drug: Placebo
- Radioactive Tablet (Part 2 only) (Other): oral radioactive tablet for scintigraphic analysis
  Interventions: Other: Radioactive Tablet (Part 2 Only)

INTERVENTIONS:
Drug: AMT-126 — Single or daily dosing at doses A, B, C, D, E, F; G, H, and I
  Other Names: no other name applicable
  Arms: AMT-126
Drug: Placebo — Single or daily dosing at doses A, B, C, D, E, F; G,H, and I
  Other Names: no other name applicable
  Arms: Placebo
Other: Radioactive Tablet (Part 2 Only) — Single dose in two periods in Part 2 (optional)
  Other Names: no other name applicable
  Arms: Radioactive Tablet (Part 2 only)

SUMMARY:
Phase 1 Study of the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of AMT-126 and Optional Pharmacoscintigraphic Assessment of Oral AMT-126

DETAILED DESCRIPTION:
A Phase 1 Study in up to 2 Parts, to Assess the Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of AMT-126 in the Fasted State (in Part 1) and to Evaluate the In Vivo Performance of an AMT-126 Oral Tablet Through Pharmacoscintigraphic Assessment in the Fed and Fasted State (in Optional Part 2) in Healthy Male and Female Subjects

ELIGIBILITY:
PART 1 & 2 (Healthy Volunteers)

Inclusion Criteria:

* Healthy male subjects and female subjects of NOCBP.
* Between 18 and 55 years of age (Part 1) and 30 and 55 years of age (Part 2), inclusive.
* A body mass index of between 18.0 and 32.0 kg/m2, inclusive.
* Contraception requirements for male & female subjects.

Exclusion Criteria:

* Known hypersensitivity or allergy to AMT-126 or excipient contained in the drug formulation.
* Clinically significant abnormalities in laboratory test results (including complete blood count, chemistry panel including kidney panel, and urinalysis).
* Presence, or history of clinically significant disease which requires treatment, as judged by the investigator.
* Evidence of current SARS-CoV-2 or COVID infection.
* Women of child-bearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent adverse events (safety and tolerability) | 5 days
  Single ascending doses of AMT-126 in healthy adult volunteers by evaluation of incidence of treatment-related adverse events as assessed by CTCAE v5.0
To assess the in vivo performance of an AMT-126 tablet formulation (Optional, Part 2 only) | 5 days
  Qualitative scintigraphic data will be compiled using the following data points for analysis: tablet release (hh:mm), location of tablet release (anatomical location), gastric emptying and arrival times (hh:mm)

SECONDARY OUTCOMES:
To assess pharmacokinetics of AMT-126 in healthy volunteers | 5 days
  Assess PK parameters (i.e. Cmax) as applicable for AMT-126

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No